CLINICAL TRIAL: NCT00431015
Title: A Phase I/II Study to Investigate the Safety, Tolerability and Potential Activity of IPI-504 in Relapsed and / or Refractory Stage IIIb (With Malignant Pleural or Pericardial Effusion), or Stage IV NSCLC Patients
Brief Title: Phase I/II Safety Study of IPI-504 in Relapsed/Refractory Stage IIIb, or Stage IV Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Infinity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPI-504-03
Record Dates: First submitted 2007-01-31; First posted 2007-02-02 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Cancer of the lung; Non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — tanespimycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: IPI-504 — IV Hsp90 inhibitor

SUMMARY:
The purpose of this study is to determine the safety, tolerability and maximum tolerated dose of IPI-504 in patients with non-small cell lung cancer (NSCLC). The study will examine how IPI-504 is absorbed, distributed, metabolized and eliminated by the body. The study will also evaluate the anti-tumor activity of IPI-504.

DETAILED DESCRIPTION:
IPI-504 is a novel small molecule inhibitor of heat shock protein 90 (Hsp90), an emerging and recently identified target for cancer therapy. Hsp90 is a protein chaperone that plays a central role in maintaining the proper folding, function and viability of various "client proteins". Many of the client proteins stabilized by Hsp90 are oncoproteins and cell-signaling proteins important in cancer cell proliferation and cancer cell survival. This clinical trial will study the effects of IPI-504 in a molecularly defined sub-group of patients who carry client proteins found in non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of a Stage IIIb (with malignant pleural or pericardial effusion) or Stage IV NSCLC
* Measurable disease by RECIST criteria.

Exclusion Criteria:

* Treatment for NSCLC with any approved or investigational product within 2 weeks of the start of IPI-504 treatment for any small molecule therapy; within 4 weeks of the start of IPI-504 treatment for any biologic or any conventional chemotherapy.
* Inadequate hematologic or renal or hepatic function
* Previous treatment with 17-AAG, DMAG or other known Hsp90 inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2007-01; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Determine potential anti-tumor activity of IPI-504 in molecularly defined sub-groups of patients by RECIST criteria | Every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lecia Sequist, MD, Principal Investigator — Massachusetts General Hospital
Locations (11):
- United States (11):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Mount Sinai Comprehensive Cancer Center, Miami, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Medical College of Georgia, Augusta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mary Crowley Cancer Research Centers - Medical City, Dallas, Texas
  - Mary Crowley Cancer Research Centers - Baylor, Dallas, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington